CLINICAL TRIAL: NCT07288047
Title: Virtual Reality as an Adjunctive Agent for the Management of Pain and Anxiety During First Trimester Procedural Abortion: a Randomized Controlled Trial
Brief Title: Virtual Reality as a Method for Pain and Anxiety Control During First Trimester Procedural Abortion
Acronym: CALM-VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Study Investigator (Other)
Responsible Party: Sponsor-Investigator, Study Investigator, Fellow, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25090152
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Abortion, First Trimester; Pain Management; Pain After Surgery; Satisfaction; Satisfaction With Care; Anxiety After Surgery
Keywords: satisfaction; virtual reality; procedural abortion; pain control; anxiety control
MeSH Terms: conditions — Agnosia; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Usual care only (Active Comparator): Usual care for pain and anxiety management during a first trimester procedural abortion includes oral ibuprofen, intracervical block, and verbal analgesia.
  Interventions: Other: Usual Care
- VR headset (Experimental): Participants will wear the VR headset during the first trimester procedural abortion, in addition to usual care for pain and anxiety management. The headset will display a meditative nature video throughout the procedure.
  Interventions: Device: VR headset; Other: Usual Care

INTERVENTIONS:
Device: VR headset — VR Headset: Meta Quest 3S Meditative nature videos provided via "Guided Meditation VR" app.
  Arms: VR headset
Other: Usual Care — Usual care for pain and anxiety management during a first trimester procedural abortion includes oral ibuprofen, intracervical block, and verbal analgesia.
  Other Names: Routine care

SUMMARY:
The goal of this clinical trial is to learn whether use of a virtual reality (VR) headset showing a meditative nature video will help reduce pain and anxiety during a first trimester procedural abortion. Investigators will enroll 72 patients undergoing a first trimester procedural abortion with usual care to manage pain and anxiety compared to use of a VR headset in addition to usual care to see if use of the VR headset will decrease pain and anxiety and increase satisfaction with the procedure.

DETAILED DESCRIPTION:
While procedural abortions are common outpatient procedures, providing optimal pain and anxiety relief during these procedures is challenging. With rapidly developing technological advances, virtual reality (VR) has emerged as a promising modality to help manage pain and anxiety control in the medical field, including obstetrics and gynecology. However, there are no studies evaluating the effect of VR on pain during a procedural abortion.

The goal of this randomized controlled trial is to primarily evaluate whether using a VR headset to display a meditative nature video as a noninvasive, low risk technology may reduce pain and anxiety for patients undergoing a first trimester procedural abortion in an outpatient setting. Investigators will also evaluate factors influencing satisfaction with the procedure. Investigators will compare use of the VR headset with usual care, to usual care only; for a first trimester procedural abortion, usual care includes oral pain medications, local anesthetic medication in the cervix, and verbal reassurance. Participants will be asked to complete a survey before, after, and one week following the procedure to assess pain, anxiety, and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Planned Parenthood of Western Pennsylvania who have decided to undergo and are eligible for a procedural abortion.
* 18 years old or older
* <14 weeks gestation on day of abortion
* Able to comprehend written English
* Willing to comply with the study protocol
* Willing and able to provide informed consent

Exclusion Criteria:

* History of vertigo
* History of epilepsy
* Claustrophobia
* Significant hearing or visual impairments (such as deafness or blindness)
* Require hearing aids
* Have an implanted medical device, such as cardiac pacemaker or defibrillator
* Require misoprostol for cervical preparation
* Prior unsuccessful attempt at abortion during this pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores during a first trimester procedural abortion | Day of enrollment: immediately preprocedure and 15 minutes postprocedure.
  Pain will be measured on a visual analogue scale during and after the procedural abortion via a REDCap survey. The scale is from 0-100, with 0 being "No pain" and 100 being the "Worst pain of my life". The difference in this score (post-procedure minus pre-procedure) is what will be compared between study arms.
Anxiety scores during a first trimester procedural abortion | Day of enrollment: immediately preprocedure and 15 minutes postprocedure.
  Anxiety will be measured on a visual analogue scale during and after the procedural abortion via a REDCap survey. The scale is from 0-100, with 0 being "No anxiety or fear" and 100 being the "Worst anxiety or fear of my life". The difference in this score (post-procedure minus pre-procedure) is what will be compared between study arms.

SECONDARY OUTCOMES:
Satisfaction with the first trimester procedural abortion | Day of enrollment (immediately postprocedure) and one week after completion of the procedural abortion.
  Satisfaction will be assessed on a Likert scale using surveys administered on the day of the procedure and one week after the procedure. A score of 1 = very dissatisfied, and a score of 5 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Study Coordinator, Study Director — Univeristy of Pittsburgh
Locations (2):
- United States (2):
  - Center for Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Planned Parenthood of Western Pennsylvania, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share the data, however it is possible we may choose to share the data with other groups or individuals interested in this topic. Should we choose to share, the data will be de-identified and a data use agreement will be executed as needed.